CLINICAL TRIAL: NCT01651026
Title: Multicentered Observational Prospective Cohort Study on Multidisciplinary Treatment of Rectal Cancer
Brief Title: Multicenter Cohort Prospective Study on Multidisciplinary Treatment of Rectal Cancer
Acronym: CROSS-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: CROSS-1
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rectal cancer

SUMMARY:
The purpose of this study is to describe the diagnostic and treatment procedures employed for patients with rectal cancer in each participating center. Outcomes to treatment, costs of treatment will be described. Exploratory analyses will be done to identify factor that influence patient prognosis, as well as factors that predict patient response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis rectal carcinoma
* Signed informed consent

Exclusion Criteria:

* Refusal or incapability of providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients at participating Institutes with confirmed diagnosis of colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-01; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
list of diagnostic procedures used in clinical practice, according to participating Institute | 5 years

OTHER OUTCOMES:
all treatments received for colorectal cancer (surgery, radiation therapy, chemotherapy, supportive care, etc) per patient | 5 years
rectal cancer surgical interventions/approaches per participating center | 5 years
disease outcomes per patient per treatment received | 5 years
estimated costs per treatment pattern per center | 5 years
factors that influence patient prognosis | 5 years
  exploratory analyses
predictive factors for response to treatment | 5 years
  exploratory analyses

CONTACTS AND LOCATIONS:
Overall Officials: G. Romano, M.D., Principal Investigator — National Cancer Institute, Naples; C. Sassaroli, M.D., Principal Investigator — National Cancer Institute, Naples; M. C. Piccirillo, M.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples
Locations (3):
- Italy (3):
  - A.O.R.N. V. Monaldi, Napoli
  - A.O.U. Federico II, Napoli
  - Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Entero-proctologico, Napoli